CLINICAL TRIAL: NCT06627231
Title: A Phase 1 Open-Label Mass Balance Clinical Trial to Investigate the Absorption, Metabolism, and Excretion of Single Oral Administration of [14C]-TEV-56286 Following Multiple Oral Administrations of Nonlabeled TEV-56286 to Healthy Male Participants
Brief Title: Mass Balance Clinical Trial With TEV-56286
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV56286-MB-10193
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEV-56286 (Experimental)
  Interventions: Drug: TEV-56286; Drug: [14C]-TEV-56286

INTERVENTIONS:
Drug: TEV-56286 — Oral capsule
  Other Names: emrusolmin
Drug: [14C]-TEV-56286 — Oral capsule
  Other Names: emrusolmin

SUMMARY:
Mass balance clinical trial with TEV-56286

DETAILED DESCRIPTION:
Primary objectives:

* To investigate the mass balance and excretion of TEV-56286 following a single oral dose of [14C]-TEV-56286
* To assess the pharmacokinetics following a single oral dose of [14C]-TEV-56286

Secondary objective:

- To evaluate the safety and tolerability of TEV-56286 following once daily multiple oral dose administration

The total duration of the clinical trial for each participant is expected to be approximately 59 days.

ELIGIBILITY:
Inclusion Criteria:

* No major trauma or surgery in the 2 months before screening or at any time between screening and the first dose of the study drug, or surgery scheduled during the clinical trial including the follow-up period.
* No history of malignancy or treatment of malignancy in the last 5 years.
* No personal or family history of arrhythmia, sudden unexplained death at a young age (before 40 years) in a first-degree relative, or long QT syndrome, or a personal history of syncope of undetermined reason or previous treatment for high blood pressure.

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* History of relevant drug and/or food allergies.
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), during work, or during participation in a clinical trial in the period of 1 year prior to screening.

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Cumulative Amount of Total Radioactivity (TRA) | Up to Day 22
Cumulative Percent of TRA From the Total Radioactive Dose Administered | Up to Day 22
Maximum Observed Plasma Concentration (Cmax) | Up to Day 22
Time to Attain Maximum Observed Plasma Concentration (Tmax) | Up to Day 22
Area Under the Plasma Concentration-time Curve up to 24 Hours Postdose (AUC0-24) | Up to Day 22
Area Under the Plasma Concentration-time Curve Up To Time t, Where t is the Last Point with Concentrations Above the Lower Limit of Quantification (AUC0-t) | Up to Day 22
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-∞) | Up to Day 22
Terminal elimination half-life (t1/2) | Up to Day 22

SECONDARY OUTCOMES:
Number of Participants With At Least One Treatment-Emergent Adverse Event | Up to Day 59
Number of Participants Who Did Not Complete the Trial Due to an Adverse Event | Up to Day 59

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site 38189, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit www.clinicalstudydatarequest.com to make your request.